CLINICAL TRIAL: NCT06352164
Title: Predicting the Clinical Efficacy of Acupuncture for Abdominal Pain in Patients With Crohn's Disease Based on Gut Microbiology and Machine Learning
Brief Title: Efficacy Classification Prediction of the Effects of Acupuncture on Abdominal Pain in Patients With Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ZYS2024-03
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; Intestinal flora; Abdominal pain; Machine learning
MeSH Terms: conditions — Crohn Disease; Abdominal Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acupuncture group (Experimental): Subjects receiving acupuncture and moxibustion treatment.
  Interventions: Other: Acupuncture treatment

INTERVENTIONS:
Other: Acupuncture treatment — The investigators selected acupoints including Zhongwan (CV12) and bilateral Shangjuxu (ST37), Sanyinjiao (SP6), Gongsun (SP4), Taichong (LR3), Taixi (KI3), Hegu (LI4), and Quchi (LI11)17 according to the World Health Organization standard. Single-use 0.30×40 mm or 0.30×25 mm acupuncture needles (Hwato, Suzhou, China) were vertically inserted into each acupoint to 20-30 mm depth to obtain a deqi sensation (a soreness, distention, numbness or heaviness sensation). Bilateral Zusanli (ST36) and Tianshu (ST25) were selected for moxibustion. Pure moxa sticks (diameter: 2.8 cm; Hanyi, Nanyang, China) were ignited and fixed on a moxibustion stand at a distance of 3-5 cm to the surface of acupoints. The temperature of skin surface at the acupoints was maintained at 43 ± 1°C and monitored with a miniature infrared thermometer (Fluke 62, Fluke Corporation, Everett, WA, USA). Acupuncture and moxibustion were concomitantly performed for 30 min.

SUMMARY:
Machine learning algorithms are applied to discover gut flora markers that predict the clinical efficacy of acupuncture, so as to screen the appropriate population for acupuncture and optimise the allocation of healthcare resources.

DETAILED DESCRIPTION:
Crohn's disease is an intestinal inflammatory disease,causing abdominal pain, diarrhea and other symptoms.The intestinal flora disorder is closely related to the occurrence and development of Crohn's disease. Acupuncture can induce remission of Crohn's disease during mild to moderate active period, improve clinical symptoms such as abdominal pain. Acupuncture can affect the gut microbiota. The aim of this study was to apply gut microbiological data and clinical data from subjects at baseline to predict the clinical efficacy of acupuncture by machine learning algorithms, and to classify patients as effective/ineffective in order to screen for suitable subjects for acupuncture.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-75, no gender limit;
2. disease in mild and moderate active period: 150≤CDAI<450 and meet at least one of the following: Serum C-reactive protein level≥5mg/L, Fecal calprotectin concentration≥250μg/g or endoscopic examination shows ulcers. remission period: CDAI <150 and meet at least one of the following: Serum C-reactive protein level<5 mg/L, Fecal calprotectin concentration <250μg/g or endoscopic examination shows no ulcer;
3. patients were not taking medication or were only taking one or more of the following drugs: mesalazine (≤4g/d and mesalazine was used for at least 1 month), prednisone (≤15mg/d and prednisone was used for at least 1 month) and / or azathioprine (≤1mg/kg/d and azathioprine was used for at least 3 month);
4. those who have not used biologics within 3 months before entering the study;
5. those who have never experienced acupuncture;
6. those who understand and agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

1. patients who are recently pregnant or in pregnancy or lactation;
2. patients with serious organic diseases;
3. patients diagnosed as psychosis;
4. patients who suffer from multiple diseases and need to take other drugs for a long time, and may affect the observation of the efficacy of this trial;
5. severe skin diseases (such as erythema nodosum, pyoderma gangrenosum, etc.), eye diseases (such as iritis, uveitis, etc.), thromboembolic diseases and other serious extraintestinal manifestations;
6. there are serious intestinal fistula, abdominal abscess, intestinal stenosis and obstruction, perianal abscess, gastrointestinal hemorrhage, intestinal perforation and other complications;
7. patients with short bowel syndrome who have undergone abdominal or gastrointestinal surgery in the past half a year;
8. there are skin diseases or defects in the selected area of acupuncture and moxibustion that cannot be performed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Characterisation of gut microflora strains predictive of acupuncture efficacy | Week 12
  Application of machine learning algorithms to discover gut microbial markers (Characterisation of intestinal flora strains) predicting clinical efficacy of acupuncture to screen for appropriate acupuncture populations.
  Criteria for judging the efficacy of acupuncture: At 12 weeks, patients had complete remission of abdominal pain ( VAS score or frequency of abdominal pain per week = 0) or remission of abdominal pain ( the reduction of VAS score or the frequency of abdominal pain ≥ 3 compare with baseline) were considered effective. Otherwise, it was considered ineffective.
  Visual Analogue Scale(VAS score):The maximum score is 0, and the minimum score is 10.Higher scores represent a greater degree of abdominal pain and higher scores mean a worse outcome.
  Frequency of abdominal pain：The maximum score is 0, and the minimum score is 7. Higher scores represent a greater degree of abdominal pain and higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Wu Huangan, PhD,MD, Study Chair — Shanghai Institute of Acupuncture, Moxibustion and Meridian
Locations (1):
- Shanghai Institute of Acupuncture, Moxibustion and Meridian, Shanghai, China

IPD SHARING:
Plan to Share IPD: No